CLINICAL TRIAL: NCT05774756
Title: A Phase 3, Double Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Setmelanotide in Patients With Acquired Hypothalamic Obesity
Brief Title: A Trial of Setmelanotide in Acquired Hypothalamic Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-493-040
Record Dates: First submitted 2023-03-01; First posted 2023-03-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Hypothalamic Obesity
Keywords: melancortin 4 receptor, MC4R
MeSH Terms: conditions — Sexual Infantilism | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Setemelanotide (Experimental): Randomized 2:1 (Setmelanotide: Placebo)
  Interventions: Drug: Setmelanotide
- Placebo (Placebo Comparator): Randomized 2:1 (Setmelanotide: Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide — Solution for daily subcutaneous injection
  Other Names: RM-493; Imcivree
  Arms: Setemelanotide
Drug: Placebo — Placebo matched to setmelanotide for daily subcutaneous injection
  Arms: Placebo

SUMMARY:
The goal of this trial is to learn how well Setmelanotide works to improve weight reduction, hunger, and quality of life in patients 4 years of age and older with acquired Hypothalamic Obesity (HO). To determine how well setmelanotide works and how safe it is, patients with HO will take a daily injection of either setmelanotide or placebo and complete trial assessments for 52 weeks on a therapeutic regimen.

A separate sub-study in patients with congenital HO is detailed under NCT06760546.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented evidence of acquired hypothalamic obesity (HO)
2. Age 4 years and older
3. Weight gain associated with the hypothalamic injury and a BMI of ≥30 kg/m2 for patients ≥18 years of age or BMI ≥95th percentile for age and sex for patients 4 to <18 years of age
4. Agree to use a highly effective form of contraception throughout the study and for 90 days after the study

Key Exclusion Criteria:

1. Diagnosis of Prader-Willi syndrome (PWS) or Rapid-onset obesity with hypoventilation, hypothalamic, autonomic dysregulation, neuroendocrine tumor syndrome (ROHHADNET)
2. Weight loss >2% in the previous 3 months for patients aged ≥18 years or >2% reduction in BMI for patients aged 4 to <18 years
3. Bariatric surgery or procedure within last 2 years
4. Diagnosis of severe psychiatric disorders; any suicidal ideation, attempt or behavior
5. Current, clinically significant pulmonary, cardiac, metabolic, or oncologic disease
6. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions (excluding non-invasive basal or squamous cell lesion)
7. History or close family history of skin cancer or melanoma
8. Participation in any clinical trial with an investigational drug/device within 3 months prior to the first trial dose
9. Previously enrolled in a clinical trial involving setmelanotide or any previous exposure to setmelanotide
10. Inability to comply with once daily (QD) injection regimen
11. If female, pregnant and/or breastfeeding
12. Patients with obesity attributable to other genetic or syndromic conditions (eg, PPL [POMC, PCSK1, LEPR, collectively], BBS) prior to the hypothalamic injury.
13. If receiving hormone replacement therapy, dose has remained stable for at least 2 months before Screening

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Mean % change in BMI | From Baseline after 52 weeks on a therapeutic regimen

SECONDARY OUTCOMES:
Proportion of patients with ≥5% reduction in BMI in adult patients (≥18 years of age) or a BMI Z-score reduction of ≥0.2 points in pediatric patients (<18 years of age) | From Baseline after 52 weeks on a therapeutic regimen
Mean change in the weekly average of the daily most hunger score in patients ≥12 years old | From Baseline after 52 weeks on a therapeutic regimen
Proportion of patients with a ≥2 point reduction in the weekly average of the daily most hunger score | From Baseline after 52 weeks on a therapeutic regimen
Mean change in Symptoms of Hyperphagia total score | From Baseline after 52 weeks on a therapeutic regimen
Proportion of patients with a ≥10% reduction in BMI | From Baseline after 52 weeks on a therapeutic regimen
Mean percent change in weight in patients ≥18 years | From Baseline after 52 weeks on a therapeutic regimen
Mean BMI-z score and BMI percentile reduction in patients <18 (using combined height and weight to report BMI in kg/m2) | From Baseline after 52 weeks on a therapeutic regimen
Proportion of patients aged ≥4 to <18 years with ≥0.2-point reduction of BMI Z-score | From Baseline after 52 weeks on a therapeutic regimen
Proportion of patients with BMI <30 kg/m2 (patients aged ≥18 years) or <95th percentile (patients aged <18 years) | From Baseline after 52 weeks on a therapeutic regimen
Mean change in physical functioning score and total score for the Impact of Weight on Quality of Life-Lite (IWQOL) | From Baseline after 52 weeks on a therapeutic regimen
Safety and tolerability of setmelanotide compared to placebo assessed by frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline after 52 weeks on a therapeutic regimen

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (28):
- United States (16):
  - UAN Pediatric Endocrinology, Birmingham, Alabama
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - University of Iowa Stead Family Department of Pediatrics, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Minnesota, Saint Paul, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Ohio State Wexner Medical Center, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Seattle Children's Hospital, Research and Foundation - Center for Integrative Brain Research, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada
- Germany (4):
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) - Ambulanzzentrum des UKE GmbH, Hamburg
  - Medicover Neuroendokrinologie, München
  - University Children's Hospital, Klinikum Oldenburg, Oldenburg
  - Universitaetsklinikum Ulm - Klinik fuer Kinder- und Jugendmedizin, Ulm
- Japan (3):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Nagano Children's Hospital, Azumino, Nagano
  - Toranomon Hospital, Minato, Tokyo
- Prinses Maxima Center for Pediatric Oncology, Utrecht, Netherlands
- United Kingdom (3):
  - Birmingham Women and Children's Hospital NHS Trust, Birmingham
  - Hull University Teaching Hospital, Hull
  - UCL Great Ormond Street Institute of Child Health, London

IPD SHARING:
Plan to Share IPD: No